CLINICAL TRIAL: NCT03758716
Title: An Open-Labeled Exploratory Study to Evaluate Safety and Efficacy of FB825 in Adults With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fountain Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FB825CLIIS-01-AD
Record Dates: First submitted 2018-11-25; First posted 2018-11-29 (Actual); Results first posted 2021-03-15 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FB825 (Experimental): Only one arm in the study. The subjects are planned to be dosed by IV injection with experimental drug FB825. The other name of FB825 is FB825-15D11, or Anti-CemX.
  Interventions: Drug: FB825, FB825-15D11, Anti-CemX

INTERVENTIONS:
Drug: FB825, FB825-15D11, Anti-CemX — Pharmaceutical form: 20mg/ml solution Route of administration: IV
  Other Names: FB825-15D11, Lot # 16-2056

SUMMARY:
The purpose of this study is to evaluate the Safety and Efficacy of FB825 in Adults with Atopic Dermatitis

DETAILED DESCRIPTION:
This is an open-labeled exploratory study to evaluate safety and efficacy of FB825 in adults with atopic dermatitis (AD). The study will be conduct at one medical center in Taiwan.

Approximately 12 subjects with atopic dermatitis (AD), who meet the criteria for study entry, will be enrolled to the one-arm-study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 20 and 65 years of age, inclusive.
2. The subject has a physician-confirmed diagnosis of chronic atopic dermatitis based on 3 years history of symptoms defined by the Eichenfield revised criteria of Hannifin and Rajka and supported by positive allergen-specific IgE at the screening visit.
3. Eczema Area and Severity Index (EASI) score ≧14 at the screening and baseline visits.
4. Investigator's Global Assessment (IGA) score ≧ 3 (5-point scale) at the screening and baseline visits.
5. ≧10 % body surface area (BSA) of AD involvement at the screening and baseline visits.

Exclusion Criteria:

1. Female subjects who are pregnant or lactating.
2. The subject is on diet or with poor intake.
3. The subject has a history of heart arrhythmias (any clinically relevant).
4. The subject has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 and 2 antibodies at screening.
5. The subject has a history of alcohol or drug abuse that would impair or risk the patients' full participation in the study, in the opinion of the investigator.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Yu Chu, MD-PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FB825
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FB825
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.75 (6.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 12
Total IgE [Mean (Standard Deviation); unit: IU/mL] — Total IgE (immunoglobulin E)
  IU/mL | 6611.53 (6693.41)
EASI Scores [Mean (Standard Deviation); unit: units on a scale] — EASI measurement follow the normal by Principal Investigator. range from 0-72. The lower the scores the better situation of the patient.
  units on a scale | 25.98 (8.34)

OUTCOME MEASURES:

1. Primary Outcome: % Change From Baseline in Total IgE
Description: Detect total IgE in serum by ImmunoCAP.
Time Frame: Day 169
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FB825
Number analyzed (Participants) | 12
percentage change | -45.57 (21.27)

2. Primary Outcome: % Change From Baseline in Allergen-specific IgE
Description: Detect specific IgE in serum by ImmunoCAP. (ex. Ragweed)
Time Frame: Day 169
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FB825
Number analyzed (Participants) | 12
percentage change | -50.16 (23.61)

3. Secondary Outcome: Change From Baseline in Total IgE
Description: Detect total IgE in serum by ImmunoCAP.
Time Frame: Day 8, 15, 29, 57, and day 85 (And Day 92, 99, 113, 141 and 169 if received the second dose of FB825)
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | FB825
Number analyzed (Participants) | 12
IU/mL
  Dose 1 Day 8 | 482.93 (1528.32)
  Dose 1 Day 15 | -137.70 (1634.09)
  Dose 1 Day 29 | -298.07 (1874.70)
  Dose 1 Day 57 | -862.73 (1934.82)
  Dose 2 Day 85 | -1956.86 (2880.48)
  Dose 2 Day 92 | -1581.65 (2253.79)
  Dose 2 Day 99 | -1419.49 (2901.00)
  Dose 2 Day 113 | -1968.97 (2668.47)
  Dose 2 Day 141 | -2350.48 (3023.13)
  Dose 2 Day 169/ EOS (end of study) | -2817.01 (3708.34)

4. Secondary Outcome: % Change From Baseline in Allergen-specific IgE
Description: Detect specific IgE in serum by ImmunoCAP. (Dog dander)
Time Frame: Day 8, 15, 29, 57, and day 85 (And Day 92, 99, 113, 141 and 169 if received the second dose of FB825)
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FB825
Number analyzed (Participants) | 12
percentage change
  Dose 1 Day 8 | -1.88 (12.87)
  Dose 1 Day 15 | -5.81 (17.92)
  Dose 1 Day 29 | -4.83 (21.74)
  Dose 1 Day 57 | -22.38 (20.98)
  Dose 2 Day 85 | -25.44 (15.01)
  Dose 2 Day 92 | -33.22 (17.42)
  Dose 2 Day 99 | -36.30 (17.80)
  Dose 2 Day 113 | -35.02 (16.81)
  Dose 2 Day 141 | -44.07 (16.40)
  Dose 2 Day 169/ EOS | -46.94 (15.02)

5. Secondary Outcome: % Changes From Baseline in Irritability Visual Analogue Scale (VAS)
Description: VAS measurement follow the normal by Principal Investigator, range from 0-20. The lower the scores the better situation of the patient.
Time Frame: Days 85
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FB825
Number analyzed (Participants) | 12
percentage change | -32.57 (30.23)

6. Secondary Outcome: % Changes From Baseline in Eczema Area and Severity Index (EASI)
Description: EASI measurement follow the normal by Principal Investigator. range from 0-72. The lower the scores the better situation of the patient.
Time Frame: Day 85
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FB825
Number analyzed (Participants) | 12
percentage change | -44.33 (41.88)

7. Secondary Outcome: % Changes From Baseline in Severity Scoring of Atopic Dermatitis Index (SCORAD)
Description: SCORAD measurement follow the normal by Principal Investigator, range from 0-103. The lower the scores the better situation of the patient.
Time Frame: Days 169
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FB825
Number analyzed (Participants) | 12
percentage change | -56.19 (15.72)

8. Secondary Outcome: % Changes From Baseline in Investigator Global Assessment (IGA) for Atopic Dermatitis
Description: IGA measurement follow the normal by Principal Investigator, range from 0-4. The lower the scores the better situation of the patient.
Time Frame: Days 169
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FB825
Number analyzed (Participants) | 12
percentage change | -39.58 (19.50)

9. Secondary Outcome: % Changes From Baseline in Body Surface Area (BSA) Involved in Atopic Dermatitis
Description: BSA measurement follow the normal by Principal Investigator, range from 0-100. The lower the scores the better situation of the patient.
Time Frame: Days 169
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FB825
Number analyzed (Participants) | 12
percentage change | -60.04 (26.41)

10. Secondary Outcome: Safety Will be Assessed by Monitoring and Recording of Adverse Events (AEs) and Serious Adverse Event (SAEs)
Description: Safety will be assessed by monitoring and recording of adverse events (AEs) and serious adverse event (SAEs); physical examination findings and vital sign measurements (systolic and diastolic blood pressures, heart rate, respiratory rate, and body temperature), clinical laboratory test results (hematology, coagulation, serum chemistry [including liver function tests, blood glucose level], and urinalysis); 12-lead ECG results.
Time Frame: through study completion, an average of 1 year.
Reporting Status: Not Posted

11. Secondary Outcome: % Changes From Baseline in Eczema Area and Severity Index (EASI)
Description: as for outcome 6
Time Frame: Day 57
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FB825
Number analyzed (Participants) | 12
percentage change | -68.09 (29.35)

12. Secondary Outcome: % Changes From Baseline in Eczema Area and Severity Index (EASI)
Description: as for outcome 6
Time Frame: Day 113
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FB825
Number analyzed (Participants) | 12
percentage change | -70.00 (34.20)

13. Secondary Outcome: % Changes From Baseline in Eczema Area and Severity Index (EASI)
Description: as for outcome 6
Time Frame: Day 141
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FB825
Number analyzed (Participants) | 12
percentage change | -73.12 (25.32)

14. Secondary Outcome: % Changes From Baseline in Eczema Area and Severity Index (EASI)
Description: as for outcome 6
Time Frame: Day 169
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | FB825
Number analyzed (Participants) | 12
percentage change | -72.14 (20.24)

ADVERSE EVENTS:
Time Frame: 169 days
Arm/Group | FB825
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 9/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FB825 (N=12)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Herpes simplex (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT03758716/Prot_SAP_000.pdf